CLINICAL TRIAL: NCT05517291
Title: Paclitaxel Coated Balloon Angioplasty Versus Primary Selective Stenting in the Treatment of TASC C/D Chronic Femoropopliteal Artery Occlusive Disease: A Multicenter Randomized Clinical Trial
Brief Title: DCB Versus Primary Selective Stenting in TASC C/D Femoropopliteal Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PASS
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Safety Issues; Efficacy, Self

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB (Experimental): participants in this group will be received drug-coated balloon angioplasty
  Interventions: Device: paclitaxel-coated balloon angioplasty or bare mental stents implantation
- stenting (Active Comparator): participants in this group will be received primary selective stenting
  Interventions: Device: paclitaxel-coated balloon angioplasty or bare mental stents implantation

INTERVENTIONS:
Device: paclitaxel-coated balloon angioplasty or bare mental stents implantation — paticipants who enrolled in this study will received paclitaxel-coated balloon angioplasty plus bailout stenting or primary bare mental stents implantation randomly

SUMMARY:
This study aims to compare the mid- and long-term outcomes between paclitaxel-coated balloon and primary selective stenting in the treatment of TASC C/D femoropopliteal artery occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 18-85yrs.
* Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved consent form.
* Subject understands the duration of the study, agrees to attend follow-up visits, and agrees to complete the required testing.
* Rutherford category 2-5.
* Subject has a de novo TASC C/D femoropopliteal artery lesions which does not exceed to the segment P1 of popliteal artery.
* The total length of target lesion ≤30cm.
* Reference vessel diameter >4 mm and <6.5 mm by visual assessment.
* Patent inflow artery with stenosis <30% and at least 1 infrapopliteal artery to the ankle (<50% diameter stenosis).
* A guidewire has successfully traversed the target treatment segment.

Exclusion Criteria:

* Acute thrombus in the target vessels.
* Vessel stenosis or occlusion due to Buerger's disease or autoimmune arteritis.
* Subject received prior stents implantation with in-stent restenosis or occlusion.
* Reintervention of the target lesion <90 days before the study procedure.
* Acquired thrombophilia or uncontrolled hypercoagulation states.
* Life expectancy <12 months.
* Severe renal（SCr≥2.5 mg/dl）or hemodialysis dependence.
* Pregnancy, suspected pregnancy, or breastfeeding during study period.
* Contraindication to contrast media or any study-required medication (antiplatelet, anticoagulant, or thrombolytic agents, etc.).
* Hypersensitivity to nitinol and/or paclitaxel.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year primary patency rate | 1 year

SECONDARY OUTCOMES:
clinical-driven target lesion revascularization | 1, 2 and 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided